CLINICAL TRIAL: NCT00005110
Title: A Multi-Centered Study of the Long-Term Effect of Salmeterol and Albuterol in Cystic Fibrosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCRR-M01RR00036-5074; M01RR000036 (NIH)
Record Dates: First submitted 2000-04-13; First posted 2000-04-14 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Salmeterol Xinafoate; Albuterol

INTERVENTIONS:
Drug: Salmeterol
Drug: Albuterol

SUMMARY:
Long term use of bronchodilators in CF is beneficial to the improvement of pulmonary function and symptoms. This study is investigating the long-term benefit of administration of the drug Salmeterol, a bronchodilator. Salmeterol will be compared to albuterol or placebo. The medication will be inhaled twice a day for 6 months.

DETAILED DESCRIPTION:
Patients that have been diagnosed with cystic fibrosis and are above 5 years and below 45 years of age are eligible. Subjects will be randomized into 1 of 3 groups. One group will get Salmeterol by multi-dose inhaler (MDI) 2 puffs 2 times a day, one group will get albuterol by MDI 2 puffs 2 times a day and the other will get placebo by MDI 2 puffs 2 times a day. Height and weight along with pulmonary function testing and vital signs will be monitored at the beginning of the study and at Visits 2, 3, and 4. Peak flow monitoring will be done each morning before study medication at home. A daily diary will be kept of this measurement. Subjects will be seen in the research center at visits 1,2,3, and 4. Telephone contact will be done at Day 15, 60, 120, and 150. Individual outcomes include a potential increase in pulmonary function testing and a decrease in frequency of pulmonary exacerbations, hospitalizations, and usage of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Ability to perform reproducible spirometry
* FEVI > 50% and < 90% (Knudsen)
* A CF pulmonary exacerbation within the last year or an FEVI<80%
* At least one delta f508 allele on CF mutation analysis
* Ability to demonstrate use of inhaled medicine and FEVI and PEFR monitor
* Written informed consent
* Negative serum pregnancy test on enrollment

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Allergy and Pulmonary Medicine, St Louis, Missouri, United States